CLINICAL TRIAL: NCT05439590
Title: The Dose-response Effect of a Four-week Intervention of Low and High Dose of Cottonseed Oil on Exercise-induced Oxidative Stress, Inflammation, and Metabolism in Healthy Adults
Brief Title: Impact of Cottonseed Oil on Oxidative Stress, Inflammation, and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cotton Incorporated 22-070
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Healthy; Oxidative Stress; Metabolic Syndrome
MeSH Terms: conditions — Inflammation; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The design is randomized parallel design, where the healthy adults will be randomized into 30 g CSO, 30 g OO, 60 g CSO, and 60 g OO.
Who Masked: Participant, Investigator
Masking Description: Smoothies containing 30 g CSO, 30 g OO, 60 g CSO, and 60 g OO were designed to be comparable in taste and appearance. The smoothies will be prepared and coded prior to receipt by the research team. Randomization is for order of coded meals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose CSO (Experimental): Participants will be randomly assigned to a smoothie containing 60 g of CSO per day for four weeks.They will be asked to consume smoothies any time of the day.
  Interventions: Behavioral: High dose CSO
- Low dose CSO (Experimental): Participants will be randomly assigned to a smoothie containing 30 g of CSO per day for four weeks.They will be asked to consume smoothies any time of the day.
  Interventions: Behavioral: Low dose CSO
- High dose OO (Active Comparator): Participants will be randomly assigned to a smoothie containing 60 g of OO per day for four weeks.They will be asked to consume smoothies any time of the day.
  Interventions: Behavioral: High dose OO
- Low dose OO (Active Comparator): Participants will be randomly assigned to a smoothie containing 30 g of OO per day for four weeks.They will be asked to consume smoothies any time of the day.
  Interventions: Behavioral: Low dose OO

INTERVENTIONS:
Behavioral: High dose CSO — Participants in the high-dose CSO arm of the study will consume two smoothies containing a total of 60 g of CSO per day for 4 weeks.
  Other Names: HD CSO
  Arms: High dose CSO
Behavioral: Low dose CSO — Participants in the low-dose CSO arm of the study will consume two smoothies containing a total of 30 g of CSO per day for 4 weeks.
  Other Names: LD CSO
  Arms: Low dose CSO
Behavioral: Low dose OO — Participants in the low-dose OO arm of the study will consume two smoothies containing a total of 30 g of OO per day for 4 weeks.
  Other Names: LD OO
  Arms: Low dose OO
Behavioral: High dose OO — Participants in the high-dose OO arm of the study will consume two smoothies containing a total of 60 g of OO per day for 4 weeks.
  Other Names: HD OO
  Arms: High dose OO

SUMMARY:
Recent research evidence suggests that cottonseed oil (CSO) may have both direct and indirect anti-inflammatory and anti-oxidative impacts linked to bioactive components of CSO and favorable alterations in lipid metabolism. These impacts are directly related to non-communicable diseases such as diabetes, cardiovascular diseases, and cancer. Our overarching hypothesis is that the effect of CSO consumption on oxidative stress markers (isoprostanes), inflammatory cytokines, metabolic biomarkers, and bile acid metabolism will be beneficial for reversing disease pathophysiology linked to oxidative stress, inflammation, and bile acids. Our long-term goal is to establish effective and practical therapeutic strategies utilizing dietary incorporation of CSO to prevent or reverse these diseases.

The following hypotheses will be tested in the proposed investigation:

H1: CSO consumption will lower exercise-induced oxidative stress, and the effect of CSO will be greater than that of OO for lowering of exercise-induced oxidative stress.

H2: CSO consumption will lower inflammatory cytokines and metabolic markers linked to the inflammation process in human participants, and the effect of CSO will be greater than that of OO for lowering inflammation.

H3: Features of serum bile acids, serum metabolomes, and lipidomes distinguishing CSO and OO treatment correspond to metabolic pathways illuminating the health benefits of CSO treatment.

H4: Metabolic and inflammatory impacts of dietary oils will be greater for 60 g/d of CSO compared to 30 g/d.

DETAILED DESCRIPTION:
The approach will be to enroll a population of healthy individuals (n=32) in a four-armed (30 g CSO, 30 g OO, 60 g CSO, and 60 g OO), randomized, double-blind, parallel controlled trial to compare the effect of these different doses of oils on exercise-induced oxidative stress.

During Visit 1, participants will undergo informed consent, anthropometric measurements, and a sub-maximal exercise test to determine their VO2max. Participants will also fill Global physical activity questionnaire (GPAQ), exercise readiness questionnaire (2022-PARQ+), AHA/ACSM Health/Fitness Facility Pre-participation Screening Questionnaire, and menstruation-related questionnaire. There will be a minimum of three days run-in periods between Visit 1 and Visit 2, during which participants will be asked to follow certain dietary guidelines such as minimal use of oil, limiting the fatty fish, omega-3, vitamin A, vitamin C, vitamin A supplements, and limiting the consumption of nuts/nut seeds/oils/oilseeds or foods containing these components. During Visit 2, participants will do an exercise test (75% VO2max for 30 mins), and a blood draw will be done before and after the exercise test. Blood will be drawn after 15 minutes of the exercise test. In addition, participants will be asked to do one month diet history questionnaire and 24 hours of dietary recall. There will be four weeks between Visit 2 and Visit 3, during which period participants will be asked to consume smoothies containing respective doses of oils every day. We will provide smoothies every week, and an additional oil will be provided in an aluminum-foil-wrapped squirt bottle for participants to substitute with their regular oil. In addition, participants will be asked to fill out a compliance check form to confirm their compliance with the study diet. There will be one weekly question on gastrointestinal issues in the compliance form. After four weeks of dietary intervention, participants will come to the lab for Visit 3. Visit 3 will follow a similar protocol to Visit 2 except that the anthropometric measurements will be done in Visit 3 as well.

Procedures:

Exercise test: During Visit 1, a sub-maximal exercise test will be done to predict how much oxygen the participant's body is able to use during exercise. This allows the researchers to have one participant exercise at the same submaximal percent of his/her maximum as all of the other participants, based on his/her fitness level. This will begin with walking on a treadmill (Woodway GmbH D79576, Weil am Rhein, Denmark) for 5 minutes at a self-selected comfortable speed at 0% grade to warm up before the test. The test involves a series of stages that get increasingly more difficult every two minutes. Participants will wear a heart rate monitor, breathe through a mouthpiece that is connected to an analyzer, and wear a nose clip. The test begins with walking, and as the participant move to more difficult stages, the intensity is increased by increasing grade and speed. The researcher will end the test when the participant has reached 85% of their age-predicted maximal heart rate (220-age in years). During visits 2 and 3, participants will report to the laboratory after an overnight fast, and blood samples will be collected before and after an exercise test. The exercise test will involve a brisk uphill walk at 75% VO2max for 30 minutes on a treadmill. During exercise, a metabolic measurement system (ParvoMedics TrueMax 2400 Metabolic System, Sandy, Utah, USA) will be used to determine a respiratory quotient and the associated level of fat oxidation. The respiratory quotient will be measured by determining the volume of carbon dioxide released over the volume of oxygen absorbed during respiration. After the blood collection, TG (and full lipid panel plus glucose) will be analyzed in real-time using a clinical chemistry analyzer (Piccolo press). At the same time, serum samples will be aliquoted and stored at -80 C until analysis for inflammatory cytokines (a profile of established mediators and biomarkers), insulin, other metabolic biomarkers linked to inflammation, and the lipidomics and metabolomics analysis. For the analysis of isoprostanes, serum samples will be snap-frozen in dry ice and ethanol slurry after it is aliquoted and immediately stored at -80 C. Investigators will measure inflammatory cytokines (TNF-α, interleukin (IL)-1β, IL-6, IL-7, IL-23, and granulocyte-macrophage colony-stimulating factor (GM-CF) using high-sensitivity Luminex multiplexing technology (Bio-Rad Bio-Plex 200 HTS) prepared by Millipore.

Dietary intervention: A registered dietitian will prepare a study diet (smoothies) which will be given to participants for four weeks. Participants will be given smoothies containing either 30 g CSO, 30 g OO, 60 g CSO, or 60 g OO per day in two separate containers. The 30 g smoothies (both CSO and OO) contain 762 kcal Calories, 120 g Carbohydrates, 3 g Protein, and 30 g Fat. The 60 g smoothies (both CSO and OO) contain 761 kcal Calories, 50 g Carbohydrates, 3 g Protein, and 30 g Fat. During these four weeks period, participants will be asked to follow certain dietary guidelines and will be asked to fill out a compliance form. Participants will be asked to fill out the compliance check form daily, indicating how much smoothie they consumed and if they consumed anything not recommended by the research team. Smoothies will be given weekly, meaning participants will visit the lab every seven days to pick up their smoothies and drop off the weekly compliance form.

Metabolomic analysis: When all samples have been collected, the serum samples will be thawed, and a metabolite fraction will be extracted. After extraction, the samples will be explored using mass spectrometry analysis. An initial targeted analysis will focus on bile acids and a set of inflammation and oxidative stress biomarkers including 8-isoPGF2a. Targeted analytes will be quantified using standard curves and the resulting concentrations will be compared using several statistical analysis tools. A deep untargeted analysis will also be undertaken which may reveal additional metabolic pathways modulated by CSO consumption. Metabolite samples will be analyzed using a Waters Synapt G2Si QTOF (Waters Corporation). This instrument has ion mobility capability and can differentiate closely related compounds, such as bile acids, in complex mixtures based on their cross-sectional area and mass. The high sensitivity and variety of scan modes make the Synapt QTOF the optimal choice for untargeted analysis of complex biological samples.

Dietary analysis: Long-term dietary habits may create adaptations that influence the response to the short-term supplementation of CSO and OO. This study will use the most recent version (2018) of the web-based Diet History Questionnaire (DHQ III), a food frequency questionnaire designed for adults 19 and older, developed by staff at the Risk Factor Monitoring and Methods Branch (RFMMB) of the NIH National Cancer Institute. The outputs of the DHQ III include carbohydrate constituents, carotenoids and tocopherols, dietary constituents from supplements, fats, fatty acids and cholesterol, macronutrients and energy, minerals, protein constituents, and vitamins are dietary constituents and food groups available in the DHQ III output files. In addition, acute dietary consumption will be determined using the free, web-based Automated Self-Administered 24-hour (ASA24®) questionnaire.

Statistical test: H1 will be tested using analysis of variance (ANOVA) to compare the differences in exercise-induced oxidative stress markers (isoprostanes) among the individuals consuming either 30 g CSO, 30g OO, or 60 g CSO, or 60 g OO. H2 will be tested using analysis of variance (ANOVA) to compare the differences in inflammation and inflammatory markers among the individuals consuming either 30 g CSO, 30g OO, 60 g CSO, or 60 g OO. To test H3, the investigator will identify changes in serum bile acids and metabolomes and then determine the metabolic pathways associated with the metabolic changes to identify potential mechanisms underlying the health impacts of CSO. To test H4, the investigator will identify the measure of serum isoprostanes, bile acids, inflammation, lipidomes, and metabolomes, and then use regression analysis to determine the level of variability in response to the different doses of CSO and OO.

ELIGIBILITY:
Inclusion Criteria:

* are between the ages of 18-55 years
* have body mass index between 18-27 kg/m2

Exclusion Criteria:

* take medications to lower cholesterol, lipids, and/or inflammation,
* take blood pressure medications,
* take antioxidant supplements (Vitamin E or C or iron) at levels greater than 800 IU/day,
* have diabetes, a gallbladder condition, or have had gallbladder removed,
* take oral contraceptives regularly,
* have smoked in the past 30 days,
* consume alcohol more than 14 drinks/week,
* have an allergy to dairy, egg, tree nuts, peanuts, shellfish, soy, fish, wheat, legumes, extra virgin olive oil, and cottonseed oil, or have been on a ketogenic or paleo diet in the past six weeks,
* pregnant or lactating,
* on weight loss diet or planning to change exercise regimen,
* have physical mobility issues or are not able to walk on a treadmill,
* or have other health concerns or conditions that may interfere with your participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Serum oxidative stress biomarkers | 4 weeks
  Concentration of exercise-induced serum isoprostanes (nM/L)
Fasting serum bile acid concentration | 4 weeks
  Concentration of fasting serum bile acids (nM/L)
Fasting serum lipids | 4 weeks
  Concentration of fasting serum triglycerides, high density lipoproteins, cholesterol, very low density cholesterol (mM)
Fasting serum inflammatory cytokines | 4 weeks
  Concentration of fasting serum inflammatory cytokine responses (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor; all in pg/ml)
Fasting serum lipidome and metabolome features (Untargeted) | 4 weeks
  Serum lipidomes and metabolomes features (Untargeted measured using LC-MS)
Fasting glucose | 4 weeks
  Serum glucose concentration (mM)
Fasting insulin | 4 weeks
  Serum insulin concentration (microIU/mL)
Fasting Eicosanoids | 4 weeks
  Several serum prostaglandins, leukotrienes, and thromboxanes (nM)

SECONDARY OUTCOMES:
Body composition | 4 weeks
  % body fat
Visceral Adipose Tissue | 4 weeks
  Quantity of adipose in liters located within the abdominal compartment
Body Mass Index | 4 weeks
  kg of body mass per meter of height squared
Blood Pressure | 4 weeks
  Systolic and Diastolic blood pressure measured in mmHg
Aerobic Fitness | 1 day
  VO2max measured in mL/kg/min

OTHER OUTCOMES:
Habitual Diet | 1 month
  Habitual dietary intake from past month reported through a food frequency questionnaire for food, beverage, and supplement intake.
Acute Diet | 1 day
  Dietary intake from the last 24-hours, self-reported through a guided online prompt
Physical activity and sedentary behavior | 7 days
  Level of physical activity and sedentary behavior measured in METminutes/week

CONTACTS AND LOCATIONS:
Overall Officials: Mary P. Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Nutrition Research Laboratory, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No